CLINICAL TRIAL: NCT03962387
Title: A Multi-center, Open, Long-term Follow-up Study to Evaluate the Efficacy and Safety of FURESTEM-AD Inj. in Patients With Moderate to Severe Chronic Atopic Dermatitis: 5-year Results From the K0102 Extension Study
Brief Title: Evalution the Safety and Efficacy in Atopic Dermatitis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: K0102-E
Record Dates: First submitted 2018-11-28; First posted 2019-05-24 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atopic Dermatitis
  Interventions: Other: Not applicable(observational study)

INTERVENTIONS:
Other: Not applicable(observational study) — Not applicable(observational study)

SUMMARY:
A multi-center, open, long-term follow-up study to evaluate the efficacy and safety of FURESTEM-AD inj. in patients with moderate to severe chronic atopic dermatitis: 5-year results from the K0102 extension study

ELIGIBILITY:
Inclusion Criteria:

1. Subject who enrolled K0102 Clinical Trial(parent study).
2. Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

1. In case follow-up is not possible from end of K0102 clinical trial to end of this study period
2. Any other condition which the investigator judges would make patient unsuitable for study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe chronic atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment (Rate of Adverse Event, Number of Participants with Adverse Event) | 5 years

SECONDARY OUTCOMES:
Percentage of subjects whose Eczema Area and Severity Index (EASI) was decreased from baseline by more than 50% at Week 12 (EASI-50) | 3 years
Percentage of subjects whose Eczema Area and Severity Index (EASI) was decreased from baseline by more than 75% at Week 12 (EASI-75) | 3 years
Rate of change in EASI from baseline | 3 years
Change in EASI from baseline | 3 years
  EASI range is from 0 (clear) to 72 (severe)
Percentage of subjects whose Investigator's Global Assessment (IGA) score at each visit is 0 or 1 | 3 years
Percentage of subjects whose IGA at each visit is 0 or 1, or improved to 2 or higher | 3 years
Percentage of subjects whose SCORing Atopic Dermatitis (SCORAD) INDEX was decreased from baseline by more than 50% at each visit (SCORAD-50) | 3 years
Rate of change in SCORAD index from baseline at each visit | 3 years
Change in SCORAD index from baseline at each visit | 3 years
  SCORAD index range is from 0 (clear) to 103 (severe)
Rate of change in Body Surface Area(BSA) of the lesion from baseline | 3 years
Change in Body Surface Area(BSA) of the lesion from baseline | 3 years
  BSA range is from 0 (clear) to 100 (severe)
Change in total serum Immunoglobulin E(IgE) from baseline | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided